CLINICAL TRIAL: NCT03153735
Title: A Multi-center, Randomized, Subject Blind, Active Controlled Design Clinical Study to Evaluate the Efficacy and Safety of CMDHA0101 as Compared to PowerFill® for Temporary Penile Enhancement
Brief Title: Clinical Study to CMDHA0101 as Compared to PowerFill® for Temporary Penile Enhancement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHA MEDITECH Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHA-CMDHA0101
Record Dates: First submitted 2017-04-05; First posted 2017-05-15 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Small Penis; Penile Enhancement
Keywords: Hyaluronic acid; Small Penis; Penile Enhancement
MeSH Terms: conditions — Penis agenesis

STUDY DESIGN:
Who Masked: Participant
Masking Description: Subject blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CMDHA0101 (Experimental): Maximum injection dose : 22 ml It is a product containing 0.3% lidocaine hydrochloride, a topical anesthetic ingredient, in a crosslinked hyaluronic acid gel
  Interventions: Device: CMDHA0101
- PowerFill® (Active Comparator): Maximum injection dose : 22 ml A white solid that was lyophilized with mixed spherical PLA (Poly-D, L-lactide) microparticles and CMC (sodium carboxymethylcellulose)
  Interventions: Device: PowerFill®

INTERVENTIONS:
Device: CMDHA0101 — Maximum injection dose : 22 ml
  Arms: CMDHA0101
Device: PowerFill® — Maximum injection dose : 22 ml
  Arms: PowerFill®

SUMMARY:
The investigators aimed to confirm the efficacy and safety of transdermal penis enlargement for 24 weeks after CMDHA0101 injection in subjects who wanted penile enlargement in male patients with small-penis syndrome *.

*Small-penis syndrome is the anxiety of thinking one's penis is too small - even though it isn't.

DETAILED DESCRIPTION:
This study was designed as a 24-week, randomized, blinded, active control trial.

If a subject signing a clinical trial agreement and satisfying the selection / exclusion criteria is enrolled in this clinical trial, he / she will receive the medical device for clinical testing at the baseline time, return to his / her home after the training . At 4 weeks, 12 weeks, and 24 weeks after the application of the medical device for clinical testing at baseline, the safety, penile girth, length, and satisfaction of the subject were evaluated. 24 weeks after application, the clinical trial sponsor (or trustee) retrieves the data necessary for the analysis of results, such as case records, for the purpose of validity and safety evaluation

ELIGIBILITY:
Inclusion Criteria:

1. Men over 20 years old and under 65 years of age
2. In screening, subjects' perception of penile size for dysmenorrhoea syndrome Those who responded with "small", "small", "normal", "large", "very large"
3. Persons who have agreed to discontinue other procedures or treatments for penile enlargement during the course of the trial
4. If the person is circumcised or has not undergone circumcision, A person who does not cover the glans
5. Those who have agreed to abstinence (sexual intercourse, masturbation, etc.) for at least one month after the medical device for clinical trial
6. Those who can understand and follow instructions
7. A person who voluntarily participates in the clinical trial and has agreed in writing to the subject consent form

Exclusion Criteria:

1. A person who has received anticoagulant or antiplatelet agent within 2 weeks before application of medical device for clinical trial or Those who need to be administered until two weeks after application (However, low-dose aspirin (300 mg / day or less) is permitted.
2. A person who has received a vitamin E preparation, NSAID preparation within 1 week of application of medical device for clinical trial or Those who need to take medicine until 1 week after application
3. Those who have a history of bleeding in past or present time
4. Persons who are adversely affected by excessive penis enlargement, which may adversely affect the operation of the medical device
5. Those who have undergone penis enlargement surgery (fat, alternative dermatologic transplantation) in the past (except for hyaluronic acid or collagen. Two years after transplantation and extension of the penis, such as suprapubic fat preparation and suspension ligament resection In the case of surgery, it is allowed.)
6. Peyronie's disease of the penis (Peyronie's disease) malformation
7. Anaphylaxis or severe allergic symptoms.

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2016-12-02 (Actual); Primary Completion 2017-11-07 (Actual); Study Completion 2017-11-07 (Actual)

PRIMARY OUTCOMES:
The difference in value from the basal value around the penis circumference after using the test device compared to the control device | baseline, 24 weeks
  Measured by value difference

SECONDARY OUTCOMES:
The difference in value from the basal value around the penis circumference after using the test device compared to the control device | baseline, 4 weeks, 12 weeks, 24 weeks
  Measured by value difference

CONTACTS AND LOCATIONS:
Overall Officials: Dae Yul Yang, Director, Study Director — Hallym University Kangdong Sacred Heart Hospital
Locations (1):
- Gangdong Sacred Heart Hospital, Hallym Univ, Seoul, Gangdong-gu/Gil-dong 445, South Korea

IPD SHARING:
Plan to Share IPD: Undecided